CLINICAL TRIAL: NCT01636999
Title: Comparing Pain Relief in Early Labor: Nitrous Oxide Versus Butorphonol Study
Brief Title: Comparing Sedara to Butorphanol in Early Labor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 12-007
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Labor Pain
Keywords: Sedara; Nitrous Oxide; Butorphanol; Visual Analog Scale
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Butorphanol (Experimental): The main study arm will be examining how well a 50% Nitrous Oxide/50% Oxygen gas mixture is in reducing labor pains in term labor patients with less than 5 cm cervical dilation, compared to 2mg of Butorphanol (a common synthetic opiod used for labor pains in this setting).
  Interventions: Drug: 50% Nitrous Oxide/50% Oxygen

INTERVENTIONS:
Drug: 50% Nitrous Oxide/50% Oxygen — The gas mixture is provided via the Sedara portable gas delivery system. This system is equipped with a non-rebreather mask which the patient holds over their mouth and nose. The delivery of the gas is only triggered by the patient's spontaneous breath. The gas machine will be provided to the patient to use as much as they like during the 60 minutes data collection period. The only dose which the machine allows to be administered is 50% Nitrous Oxide/50% oxygen.
  Other Names: Sedara (FDA 510K Approval No. K101286)

SUMMARY:
Nitrous oxide (N2O) has been used for the treatment of labor pains for over 150 years. The longevity of its use in clinical practice can be attributed to its excellent safety profile, ease of administration, and familiarity of use among health-care providers. Sedara is a self-administered 50% N2O, 50% oxygen gas mixture with pain relieving and anxiety reducing properties recently available for use in the United States (US) to treat various painful clnical situations, including labor pains.

In the US, epidural or intravenous administration of narcotic medications is one of the most common and frequently requested treatments for patients experiencing labor pains. Although generally considered safe, complications are common with epidurals, including fetal distress, low blood pressure in the mother, respiratory distress, and headache. In our hospital system, the use of the synthetic intravenous painkiller, Butorphanol, is a mainstay of treatment for labor pains. It too can have undesirable side effects in the mother, including low blood pressure and breathing problems.

Because Sedara has until recently been unavailable in the US, studies comparing its efficacy with other agents for labor pain have been confined to Europe, predominantly in the United Kingdom. Several studies have investigated the efficacy of Sedara versus inhalation and intravenous anesthetics in various countries. We have obtained several Sedara devices for use in the West Penn Allegheny Health System (WPAHS) Department of Anesthesiology and would like to examine its efficacy in our target population of women experiencing pain during early labor.

Hypothesis - Sedara will provide equivalent or superior pain relief among term, adult parturients in early labor (less than 5cm cervical dilation) compared to intravenous butorphanol.

Primary aim - Compare Sedara versus butorphanol in a single-blinded randomized trial with the main outcome measure being reduction in labor pains at various time intervals.

Our findings may be significant in terms of improving safety and efficacy of pain relief among women experienceing labor pains. Given that Sedara has not been previously studied in the US, the results may influence current obstetrical and pain management practices.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Presents in active labor
* Full term pregnancy (at least 37 and up to 42 weeks gestation)
* Less than 5 cm cervical dilation on exam

Exclusion Criteria:

* Patients who have received prior regional or opioid analgesia
* Patients who have taken oral analgesics (narcotic or non-steroidal anti inflammatory drugs) within 6 hours prior to presentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 60 minutes
  The primary outcome measure of pain relief will be measured using a 100mm visual analog scale (VAS) immediately prior to administration of the test medication (either Sedara or butorphanol) and again at 5, 15, 30 and 60 minutes following the medication start time.

SECONDARY OUTCOMES:
Nausea, Sedation, Satisfaction | 60 minutes
  Secondary outcome measures collected include maternal reported level nausea, sedation, and overall satisfaction with analgesia using the Visual Analog Scores Scale at 0, 5, 15, 30 and 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Helene Finegold, MD, Principal Investigator — Associate Residency Program Director; Christopher Troianos, MD, Study Chair — Residency Program Director
Locations (1):
- West Penn Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Volmanen P, Palomaki O, Ahonen J. Alternatives to neuraxial analgesia for labor. Curr Opin Anaesthesiol. 2011 Jun;24(3):235-41. doi: 10.1097/ACO.0b013e328345ad18. PMID 21451402
- [Background] Rosen MA. Nitrous oxide for relief of labor pain: a systematic review. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S110-26. doi: 10.1067/mob.2002.121259. PMID 12011877
- [Background] Maslekar S, Gardiner A, Hughes M, Culbert B, Duthie GS. Randomized clinical trial of Entonox versus midazolam-fentanyl sedation for colonoscopy. Br J Surg. 2009 Apr;96(4):361-8. doi: 10.1002/bjs.6467. PMID 19283736
- [Background] Young P, Emery NC, Reisin R. Epidural analgesia for labor and delivery. N Engl J Med. 2010 Jul 22;363(4):395. No abstract available. PMID 20677364
- [Background] Viscomi CM. Randomized trial of epidural versus intravenous analgesia during labor. Obstet Gynecol. 1996 Mar;87(3):480-2. doi: 10.1016/0029-7844(96)82976-0. No abstract available. PMID 8598984
- [Background] Dickinson JE, Paech MJ, McDonald SJ, Evans SF. Maternal satisfaction with childbirth and intrapartum analgesia in nulliparous labour. Aust N Z J Obstet Gynaecol. 2003 Dec;43(6):463-8. doi: 10.1046/j.0004-8666.2003.00152.x. PMID 14712952
- [Background] Yeo ST, Holdcroft A, Yentis SM, Stewart A, Bassett P. Analgesia with sevoflurane during labour: ii. Sevoflurane compared with Entonox for labour analgesia. Br J Anaesth. 2007 Jan;98(1):110-5. doi: 10.1093/bja/ael327. PMID 17158129
- [Background] Volmanen P, Akural E, Raudaskoski T, Ohtonen P, Alahuhta S. Comparison of remifentanil and nitrous oxide in labour analgesia. Acta Anaesthesiol Scand. 2005 Apr;49(4):453-8. doi: 10.1111/j.1399-6576.2005.00639.x. PMID 15777291
- [Background] Talebi H, Nourozi A, Jamilian M, Baharfar N, Eghtesadi-Araghi P. Entonox for labor pain: a randomized placebo controlled trial. Pak J Biol Sci. 2009 Sep 1;12(17):1217-21. doi: 10.3923/pjbs.2009.1217.1221. PMID 19943458
- [Background] Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov;5(11):1086-90. doi: 10.1111/j.1553-2712.1998.tb02667.x. PMID 9835471
- [Background] Yamamoto LG, Nomura JT, Sato RL, Ahern RM, Snow JL, Kuwaye TT. Minimum clinically significant VAS differences for simultaneous (paired) interval serial pain assessments. Am J Emerg Med. 2003 May;21(3):176-9. doi: 10.1016/s0735-6757(02)42255-3. PMID 12811707
- [Background] Lee JS, Hobden E, Stiell IG, Wells GA. Clinically important change in the visual analog scale after adequate pain control. Acad Emerg Med. 2003 Oct;10(10):1128-30. doi: 10.1111/j.1553-2712.2003.tb00586.x. PMID 14525749